

# Statistical Analysis Plan

NCT Number: NCT04941898

Title: ADYNOVATE SPECIAL DRUG USE RESULT SURVEY (Perioperative

Administration)

Study Number: TAK-660-5002

Document Version and Date: Original / 30-Jan-2024

Certain information within this document has been redacted (ie, specific content is masked irreversibly from view) to protect either personally identifiable information or company confidential information.

Note; This document was translated into English as the language on original version was Japanese.

# Statistical Analysis Plan

Takeda Pharmaceutical Company Limited.

Director, Biostatistics Property of Lan

Original: Prepared on January 30, 2024

# TABLE OF CONTENTS

| List of Terms and Abbreviations | 3 |
|---|---|
| Analysis Sets | 4 |
| Safety specification (Important identified risks, important potential risks, and | 3<br>4<br>5<br>6 eths |
| important missing information) | 5 |
| 1 Number of study sites and patients enrolled and patient composition | 6 |
| 1.1 Subject Disposition (Patient Disposition Chart) | 6 |
| 2. Patient characteristics | ~ 7 |
| 2.1 Patient characteristics | 7 |
| 3 Details of treatment | 9 |
| 2.1 Patient characteristics 3 Details of treatment 3.1 Surgery Performed 3.2 Intraoperative status | 9 |
| 3.2 Intraoperative status | 9 |
| 3.3 Administration status of this drug | 9 |
| 3.4 Perioperative Management Completion Status | 9 |
| 4 Matters related to safety | 11 |
| 4.1 Status of Occurrence of Adverse Events and Adverse Drug | |
| Reactions/Infections | 11 |
| 4.1.1 Occurrence of adverse events | |
| 4.1.2 Occurrence status of adverse reactions/infections | 11 |
| 4.1.3 Incident Status of Adverse Events and Adverse Drug | |
| Reactions/Infections Included in Safety Specifications | . 12 |
| 4.2 Status of occurrence of adverse events, adverse drug reactions, and | |
| infections in patients excluded from safety evaluation | . 15 |
| 4.2.1 Status of adverse events in patients excluded from safety evaluation | . 15 |
| 4.2.2 Occurrence Status of Adverse Reactions/Infections in Patients | |
| Excluded from Safety Evaluation | . 15 |
| 4.3 Occurrence Status of Adverse Events and Adverse Drug | |
| Reactions/Infections by Seriousness, Time to Onset, Outcome, and | |
| Causal Relationship with this drug | . 15 |
| 4.3.1 Occurrence of adverse events by seriousness, timing of onset, outcome | , |
| and causal relationship with this drug | . 15 |
| 4.3.2 Occurrence Status of Adverse Reactions/Infections by Seriousness, | |
| Onset Timing, and Outcome | . 17 |
| 4.4 Factors that may affect the safety | . 18 |
| 4.4.1 Onset status of adverse reactions/infections by patient background | |
| and treatment factors | . 18 |

| | 4.4.2 Occurrence Status of Adverse Reactions/Infections by Gender | 19 |
|---|---|---|
| | 5 Efficacy | 20 |
| | 5.1 hemostatic effect | 20 |
| | 6 Occurrence Status of Adverse Reactions/Infections in Additional | |
| | Pharmacovigilance Plan | 21 |
| | 6.1 Incidences of ADRs and infections included in additional | d |
| | pharmacovigilance plan (Attached Form 12) | 21 🛇 |
| | 7 Case Summary for Post-marketing Surveillance, etc | |
| | 7.1 Case summary in post-marketing surveillance, etc. (Attached Form 16) | 22 |
| | Preparation history (version control) | 23 |
| | Preparation history (version control) | 1 |
| Property | Preparation history (version control) [Appendix 1] Comparison table of changes Adda to the comparison table of changes and authority the comparison table of changes are comparison to the comparison table of changes and authority the comparison table of changes are comparison to the change and authority the comparison table of changes are comparison to the change and authority the cha | |

# List of Terms and Abbreviations

- This drug: ADYNOVATE Intravenous Kit is abbreviated as this drug.
- This statistical analysis plan uses "adverse drug reactions/infections" in the title and "adverse drug reactions" in the text and tables.

  Serious adverse events: Adverse events assessed.

  listed in the ModD.
- listed in the MedDRA code list (PT code) of the Important Medical Events List will be handled as serious even if the investigator's assessment is "non-serious."
- "Related" to this drug: Adverse events other than those "not related" to this drug will be handled as "related," and adverse events "not related" to this drug will be handled as "not related."
- Summary statistics: A collective term for sample size, mean, standard deviation, maximum, minimum, and quartiles.
- Patients whose CRFs were not collected: Registered patients whose CRFs were not collected.
- Patients whose CRFs were collected: Registered patients whose CRFs were collected.
- Timing of onset of an adverse event (or adverse drug reaction, etc.): Calculated as the date of onset of the adverse event (or adverse drug reaction, etc.) - the start date of the first dose of this drug +1.
  - If the date of onset of an adverse event (or adverse drug reaction, etc.) is unknown, it will be calculated as January 1. However, if year of initial administration of this drug = year of onset of adverse event (or adverse drug reaction), it will be calculated as month and day of initial administration of this drug.
    - If the start date of an adverse event (or adverse drug reaction) is unknown, it will be counted as day 1. However, if the date of initial administration of this drug = the date of onset of an adverse event (or adverse reaction, etc.), this will be calculated as the date of initial administration of this drug.

# **Analysis Sets**

In this survey, "patients evaluated for safety" and "patients evaluated for efficacy" will be set as analysis sets. This analysis set will be defined as follows:.

• Subjects evaluable for safety

Defined as "Patients receiving this drug who had no major protocol violations and whose safety could be evaluated." Specifically, patients with locked CRFs who meet any of the following criteria will be excluded from the safety analysis set.

- This drug not administered
- Enrollement outside the registration period
- Unknown presence/absence of adverse event
- Patients eligible for efficacy evaluation

Defined as "Patients evaluable for efficacy with no major protocol deviations among patients And the state of t evaluated for safety." Patients who meet the following conditions among the patients evaluated for safety will be excluded from the patients evaluated for efficacy.

# Safety specification (Important identified risks, important potential risks, and important Ce applicable reims of Use vity c missing information)

- Important identified risks
  - Inhibitor Development: Any of the following:.
    - PT: Factor VIII inhibition
  - PT: Anti Factor VIII antibody positive
  - PT: Antibody test positive
  - PT: Anti factor VIII antibody increased
  - SMQ: Lack of efficacy/effect (Narrow)
- Property of Takeda. For noncommercial use only and subject to Shock, anaphylaxis: Events falling under the SMQ of hypersensitivity (Narrow).

# Number of study sites and patients enrolled and patient composition

# **Subject Disposition (Patient Disposition Chart)**

Analysis All enrolled patients (patients enrolled)

population:

Analysis item: Patients enrolled

> Number of study sites CRF not collected

CRF collected

Patients excluded from safety

evaluation \*

oplicable Terms of Use ehro [this drug not administered enrollment Reason for exclusion (multiple counting) outside the registration period, unknown presence/absence of adverse events]

Subjects evaluable for safety Patients excluded from efficacy

evaluation \*

[Other than the target disease] Reason for exclusion

Patients eligible for efficacy

evaluation

Analytical method:

Property of Lakeda. For

For the above analytical variables, the following analyses will be performed to prepare the patient composition chart.

For registered patients, the number of study sites is also shown. The same medical institution with different departments in the survey shall be counted as one medical institution. If there is no subject applicable to the reason for exclusion, 0 subject is displayed. In addition, the number of cases will be displayed for "cases whose CRFs have been collected," "cases whose CRFs have not been collected," "cases subject to safety evaluation," "cases excluded from safety evaluation," "cases subject to efficacy evaluation," and "cases excluded from efficacy evaluation." For patients excluded from the safety evaluation and efficacy evaluation, the number of patients by reason for exclusion will be tabulated and listed.

\*"Patients excluded from safety evaluation" refers to locked patients who were excluded from the "patients eligible for safety evaluation." Similarly, "patients excluded from efficacy evaluation" refer to "patients excluded from efficacy evaluation" among the "patients evaluated for safety."

Frequency tabulations

### 2 **Patient characteristics**

### **Patient characteristics** 2.1

Analysis Subjects evaluable for safety

population:

Analysis item: Gender [Male, female]

> Min<= - <12, 12<= - <18, 18<= - <65, Age (years)

> > $65 \le - \le Max$

[Absent, present, unknown] Presence/absence of a history

of surgery

Presence or absence of medical [Absent, present, unknown]

history

[Hepatitis C, Hepatitis B, and others] Details of medical history

(duplicate counting)

Complications [Absent, present]

Details of complications

[Hepatitis C, hepatitis B, chronic hepatitis, (duplicate counting)

hepatic cirrhosis] Liver disease

Renal disease [Nephrotic syndrome, glomerulonephritis,

chronic renal failure]

Other diseases

Hypersensitivity predisposition [Absent, present, unknown]

Height (cm) [Min<= - <140, 140<= - <150, 150<= -

<160, 160<= - <170, 170<= - <= Max, not

measured]

Weight (kg)  $[Min \le - <50, 50 \le - <65, 65 \le - <=Max]$ 

Age at diagnosis of hemophilia [Min<= - <18, 18<= - <65, 65<= - <70,

 $70 \le - < 75, 75 \le - < 80, 80 \le - < = Max$ 

Severity of Hemophilia A [Severe, Moderate, Mild]

Family history of hemophilia A [Absent, present, unknown]

Details of family history of [Father, mother (Hemophilia A, carrier),

hemophilia A (overlapping brother/sister, grandparent, etc.]

tabulation)

Property of Takedai. For

History of FVIII inhibitor [Absent, present, unknown]

development

Presence or absence of a [Absent, present, unknown]

history of treatment with this

drug before perioperative

management

Before the start of [Absent, present, unknown]

perioperative management

(most recent)

Presence or absence of

treatment for hemophilia A

[ADYNOVATE, ADVATE, others] Before the start of

perioperative management

(most recent)

Treatment of hemophilia A

[Product name] (Multiple

counting)

[Prophylaxis, on-demand treatment, Before the start of

perioperative management

(most recent)

Treatment of hemophilia A

[Administration method]

(overlapping tabulation)

only and subi For the above analytical variables, frequency tabulation of discrete data and an statistic sta Analytical

summary statistics of continuous data will be calculated.

8

# **Details of treatment**

# **Surgery Performed** 3.1

Subjects evaluable for safety Analysis

population:

Analysis item: Type of Surgery

Analytical Frequency of the number of types of surgery will be tabulated.

method:

# 3.2 **Intraoperative status**

Subjects evaluable for safety **Analysis** 

population:

Analysis item: Intraoperative blood loss (mL)

Transfusion status

[Absent, present]
[Packed red bloo's latelets, fre-bser' Type of transfusion (duplicate counting)

Drainage [Absent, present]

[Open, semi-closed and closed drains] Drain type (duplicate counting)

For the above analytical variables, frequency tabulation of the number of Analytical

discrete data and summary statistics based on the number of continuous data method:

will be calculated for overall data, major surgery, and minor surgery.

## Administration status of this drug 3.3

Analysis Subjects evaluable for safety

population:

Duration of treatment (days) Analysis item:

Dose (IU)

Analytical

For the above analytical variables, summary statistics based on the number of events will be calculated. One form will be prepared for each preoperative,

intraoperative, and postoperative period. At that time, summary statistics will

be calculated by administration method (Bolus, continuous infusion) for

before and during surgery. For postoperative cases, summary statistics will be

calculated by administration method (Prophylaxis, continuous infusion,

others).

# Property of Lakeda **Perioperative Management Completion Status**

Subjects evaluable for safety

population:

[Due to the onset of adverse events, the patient did not visit the hospital before the completion of perioperative management, etc., due to insufficient effect, etc.]

allytical variables, frequency of the number of events will be add to the add the add to the add the add to the add the add to the add the add to the add the add to the add

10

# 4 Matters related to safety

# 4.1 Status of Occurrence of Adverse Events and Adverse Drug Reactions/Infections

# 4.1.1 Occurrence of adverse events

Analysis population: Subjects evaluable for safety

Analysis item: Adverse Events

Analytical method: For the above analytical variable, the following analyses should be

performed.

(1) Number of subjects with adverse events

(2) Number of AEs

(3) Incidence of adverse events

(4) Type of Adverse Event

The calculation method for each analysis is as follows.

[Number of subjects with adverse events]

• Number of patients with adverse events.

[Number of adverse events]

 Number of AEs that occurred. If the same adverse event occurs more than once in the same patient, the total number of events will be tabulated.

[Incidence of adverse events]

 Calculated as the number of patients with adverse events/number of patients evaluated for safety ×100.

[Type of adverse event]

- AEs will be coded using MedDRA/J. It will be roughly classified by SOC and tabulated by PT. SOC of "investigations" will be summarized by HLGT (Sort in ascending order of HLGT code, but do not output) and PT.
- Within SOC, the number of patients with adverse events and the
  incidence rate will be described using internationally agreed SOC
  order. A subject with multiple occurrences of an event within an
  SOC should be counted only once for that SOC.
- By PT, the number of patients with adverse events and the
  incidence will be described in ascending order of PT codes. A
  subject who experienced the same PT more than once should be
  counted as 1 subject with the PT.

# ated by PT a by HLGT (Sort do not output) and PT. Within SOC, the number of princidence rate will be described order. A subject with multiple SOC should be counted only By PT, the number of patient incidence will be described it subject who experienced the counted as 1 subject with the

Analysis population: Subjects evaluable for safety

Analysis item:

Adverse reactions, etc.

Analytical method:

For the above analytical variable, the following analyses should be performed.

- (1) No. of patients with adverse reactions, etc.
- (2) Adverse drug reactions, etc. Number of events
- (3) Incidence of adverse drug reactions, etc.
- (4) Adverse reactions, etc. type

The calculation method for each analysis is as follows.

[Number of patients with adverse reactions]

• Number of patients with adverse reactions, etc.

[Number of adverse reactions]

 Number of adverse drug reactions, etc. that occurred. If the same adverse drug reaction, etc. occurs multiple times in the same patient, the total number of events will be tabulated.

[Incidence of adverse reactions]

 Number of patients with adverse drug reactions/Number of patients evaluated for safety ×100.

[Types of adverse reactions, etc.]

- Adverse drug reactions will be coded using MedDRA/J. It will be roughly classified by SOC and tabulated by PT. SOC of "investigations" will be summarized by HLGT (Sort in ascending order of HLGT code, but do not output) and PT.
- In SOC, the number of patients with adverse drug reactions, etc. and the incidence will be described in SOC internationally agreed order. A subject with multiple occurrences of an event within an SOC should be counted only once for that SOC.
- By PT, the number of patients with adverse drug reactions, etc. and the incidence will be described in ascending order of PT codes. A subject who experienced the same PT more than once should be counted as 1 subject with the PT.
- 4.1.3 Incident Status of Adverse Events and Adverse Drug Reactions/Infections Included in Safety Specifications
- 4.1.3.1 Incidences of adverse events included in the safety specifications (tabulation by risk)

Analysis population: Subjects evaluable for safety

Analysis item: Adverse events corresponding to important identified risks (Inhibitor

development, shock/anaphylaxis) in the safety specifications

Stratification item: **Total** 

> Seriousness [Serious, non-serious]

Analytical method: For the above analytical variable, the following analyses should be

performed for each risk and each stratum of the stratification factor. oplicable The risks to be included are defined as described in the Safety

Specification (Important Identified Risks).

[Number of subjects with adverse events]

Number of patients with adverse events.

[Number of adverse events]

Number of AEs that occurred. If the same adverse event occurs more than once in the same patient, the total number of events will be tabulated.

[Incidence of adverse events]

Calculated as the number of patients with adverse events/number of patients evaluated for safety  $\times 100$ .

[Type of adverse event]

- AEs will be coded using MedDRA/J. It will be roughly classified by SOC and tabulated by PT. SOC of "investigations" will be summarized by HLGT (Sort in ascending order of HLGT code, but do not output) and PT.
- Within SOC, the number of patients with adverse events and the incidence rate will be described using internationally agreed SOC order. A subject with multiple occurrences of an event within an SOC should be counted only once for that SOC. However, if there are differences in the category of each stratification item, the subject will be counted as 1 subject in each category. For the last stratification item, 1 will be adopted according to the priority.
- Property of Lakeda. For non-co By PT, the number of patients with adverse events and the incidence will be described in ascending order of PT codes. A subject who experienced the same PT more than once should be counted as 1 subject with the PT. However, if there are differences in the category of each stratification item, the subject will be counted as 1 subject in each category. For the following stratification items, 1 item will be adopted in accordance with the priority order.

Seriousness: Serious → Non-serious

# Inhibitor development, shock/anaphylaxis) in the safety specifications Total Seriousness [Serious For the above analytical 4.1.3.2 Incident Status of Adverse Reactions/Infections Included in Safety Specifications (Tabulation by Risk)

Analysis population:

Analysis item:

Stratification item:

Analytical method:

performed for each risk and each stratum of the stratification factor.

The risks to be included are defined as described in the Safety

Specification (Important Identified Risks).

[Number of patients with adverse reactions]

Number of patients with adverse reactions, etc..

[Number of adverse reactions]

Number of adverse drug reactions, etc. that occurred. If the same adverse drug reaction, etc. occurred multiple times in the same patient, the total number of events will be tabulated.

[Incidence of adverse reactions]

Number of patients with adverse drug reactions/Number of patients evaluated for safety  $\times 100$ .

[Type of adverse reactions, etc.]

- Adverse drug reactions will be coded using MedDRA/J. It will be roughly classified by SOC and tabulated by PT. SOC of "investigations" will be summarized by HLGT (Sort in ascending order of HLGT code, but do not output) and PT.
- Property of Takedai. For non-co In SOC, the number of patients with adverse drug reactions, etc. and the incidence will be described in SOC internationally agreed order. A subject with multiple occurrences of an event within an SOC should be counted only once for that SOC. However, if there are differences in the category of each stratification item, the subject will be counted as 1 subject in each category. For the last stratification item, 1 will be adopted according to the priority.
  - By PT, the number of patients with adverse drug reactions, etc. and the incidence will be described in ascending order of PT codes. A subject who experienced the same PT more than once

should be counted as 1 subject with the PT. However, if there are differences in the category of each stratification item, the subject Seriousness: Serious → Non-serious

Status of occurrence of adverse events, adverse drug reactions, and infections in patients excluded from safety evaluation

Status of adverse events in patients excluded from safety evaluation

lysis population: Patients excluded from safety evaluation

ysis item: Adverse Events

ytical method: For the above analytical variables.

# 4.2

# 4.2.1 Status of adverse events in patients excluded from safety evaluation

Analysis population:

Analysis item:

Analytical method:

# 4.2.2 Occurrence Status of Adverse Reactions/Infections in Patients Excluded from **Safety Evaluation**

Patients excluded from safety evaluation Analysis population:

Adverse reactions, etc. Analysis item:

For the above analytical variable, analyses should be performed in the Analytical method:

same manner as in Section 4.1.2.

# Occurrence Status of Adverse Events and Adverse Drug Reactions/Infections by 4.3 Seriousness, Time to Onset, Outcome, and Causal Relationship with this drug

# 4.3.1 Occurrence of adverse events by seriousness, time of onset, and outcome

Analysis population: Subjects evaluable for safety

Analysis item: Adverse Events

Property of Takeda. Stratification item: Total

Seriousness [Serious, non-serious]

[1<= -<=5, 6<= -<=10, 11<= -<=20, Timing of onset (day)

 $21 \le - \le 30, 31 \le - \le Max$ 

[Recovered/resolved, resolving, not Outcome

recovered, recovered with sequelae,

fatal (due to this event), unknown]

Analytical method: For the above analysis set, the following analyses should be performed

for each stratum of the stratification factor.

(1) Number of subjects with adverse events

- (2) Number of AEs
- (3) Incidence of adverse events
- (4) Type of Adverse Event

The calculation method for each analysis is as follows.

[Number of subjects with adverse events]

Number of patients with adverse events.

[Number of adverse events]

Number of AEs that occurred. If the same adverse event occurs more than once in the same patient, the total number of events will be tabulated.

[Incidence of adverse events]

Calculated as the number of patients with adverse events/number of patients evaluated for safety ×100.

[Type of adverse event]

- AEs will be coded using MedDRAV. It will be roughly classified by SOC and tabulated by PT. SOC of "investigations" will be summarized by HLGT (Sort in ascending order of HLGT code, but do not output) and PT.
- Within SOC, the number of patients with adverse events and the incidence rate will be described using internationally agreed SOC order. A subject with multiple occurrences of an event within an SOC should be counted only once for that SOC. However, for the same SOC, 1 case shall be adopted according to the order of priority at the end.
- Property of Takedai. For nonico By PT, adverse events The number of patients with adverse events and the incidence will be described in ascending order of PT codes. A subject who experienced the same PT more than once should be counted as 1 subject with the PT. However, for the same PT, adopt 1 case in the following order of priority.

Seriousness: Serious → Non-serious

Time of onset: 1-5 days  $\rightarrow$  6-10 days  $\rightarrow$ 11 to 20 days  $\rightarrow$ 21 to 30

 $days \rightarrow \geq 31 days$ 

Outcome: Death (due to this event)  $\rightarrow$  recovered with sequelae  $\rightarrow$ 

not recovered → recovering → recovered → unknown

# 4.3.2 Occurrence Status of Adverse Reactions/Infections by Seriousness, Onset Timing, and Outcome

Analysis population: Subjects evaluable for safety

Analysis item: Adverse reactions, etc.

Stratification item: Total

Seriousness

Timing of onset (day)

Outcome

[1<= - <= 5, 6<= - <= 10, 11<= - <= 20, 21<= - <= 30, 31<= - <= Max]

[Recovered/resolved "
recovered." recovered, recovered with sequelae,

fatal (due to this event), unknown]

For the above analysis set, the following analyses should be performed Analytical method:

for each stratum of the stratification factor.

(1) No. of patients with adverse reactions, etc.

(2) Adverse drug reactions, etc. Number of events

(3) Incidence of adverse drug reactions, etc.

(4) Adverse reactions, etc. type

The calculation method for each analysis is as follows.

[Number of patients with adverse reactions]

Number of patients with adverse reactions, etc..

Number of adverse drug reactions, etc. that occurred. If the same adverse drug reaction, etc. occurred multiple times in the same patient, the total number of events will be tabulated.

Number of patients with adverse drug reactions/Number of patients evaluated for safety ×100.

- with the content of t Adverse drug reactions will be coded using MedDRA/J. It will be roughly classified by SOC and tabulated by PT. SOC of "investigations" will be summarized by HLGT (Sort in ascending order of HLGT code, but do not output) and PT.
  - In SOC, the number of patients with adverse drug reactions, etc. and the incidence will be described in SOC internationally agreed order. A subject with multiple occurrences of an event within an SOC should be counted only once for that SOC. However, for the

- same SOC, 1 case shall be adopted according to the order of priority at the end.
- Loues. A subject who experienced the same

  I more than once should be counted as 1 subject with the PT.

  However, for the same PT, adopt 1 case in the following order of priority.

  Seriousness: Serious 

  Non-serious

  Time of onset: 1-5 -1

 $days \rightarrow \geq 31 days$ 

Outcome: Death (due to this event)  $\rightarrow$  recovered with sequelae  $\rightarrow$ 

not recovered  $\rightarrow$  recovering  $\rightarrow$  recovered  $\rightarrow$  unknown

# Factors that may affect the safety

# 4.4.1 Onset status of adverse reactions/infections by patient background and treatment factors

Subjects evaluable for safety Analysis population:

Adverse reactions, etc. Analysis item:

Stratification item: Gender [Male, female]

> Age (years)  $Min \le - <12, 12 \le - <18,$

> > $18 \le -65, 65 \le -8$

Presence/absence of a history of [Absent, present, unknown]

surgery

Presence or absence of medical [Absent, present, unknown]

history

Complications [Absent, present]

Hypersensitivity predisposition [Absent, present, unknown] Severity of Hemophilia A [Severe, Moderate, Mild] History of FVIII inhibitor [Absent, present, unknown]

development

Property of Takedai. For not

Presence or absence of a history of [Absent, present, unknown]

treatment with this drug before

perioperative management

Before the start of perioperative [Absent, present, unknown]

management (most recent)

Presence or absence of treatment

for hemophilia A

Analytical method: For the above analysis set, the following analyses should be performed

for each stratum of the stratification factor.

- (1) Number of patients with adverse reactions, etc.
- (2) Incidence of adverse drug reactions

The calculation method for each analysis is as follows.

[Number of patients with adverse reactions]

Number of patients with adverse reactions, etc.

[Incidence of adverse reactions]

Number of patients with adverse drug reactions/Number of patients

4.4.2 Occurrence Status of Adverse Reactions/Infections by Age
Analysis population: Subjects evaluable for safety
Analysis item.

Stratification item:

[Min<= - <18, 18<= - <65, 65<= - <70, 70<= - <75, 75<= - <80, Age (years)

For the above analytical variable, the same analyses as those in Section Analytical method: en will be will be will be roperty of takeda. For non-commercing

4.1.2 will be performed for each stratum of the stratification factor.

# **Efficacy**

### hemostatic effect 5.1

Analysis population: Patients eligible for efficacy evaluation

Analysis item: hemostatic effect

Kerms of Use At evaluation point: During surgery, on postoperative Day 1, and at the time of completion

(or discontinuation) of postoperative perioperative management

**Evaluation Category:** [Markedly effective, effective, slightly effective, ineffective]

Abulate vents at each vents at For the above analytical variables, frequency will be tabulated for the Analytical method:

number of patients evaluated and the number of events at each

20

# Occurrence Status of Adverse Reactions/Infections in Additional Pharmacovigilance Plan

# 6.1 Incidences of ADRs and infections included in additional pharmacovigilance plan (Attached Form 12)

Analysis Subjects evaluable for safety

population:

Adverse reactions, etc. corresponding to safety specifications (Important Analysis item:

identified risks, important potential risks, and important missing information)

Seriousness Stratification [Serious, non-serious]

item:

For the above analytical variables, the following analyses should be Analytical

performed for each of the subgroups of the stratification factors in accordance method:

with (Note) 1~4 in Attached Form 12 to PSEHB/PED Notification No. 0325-

10 dated March 25, 2020.

(1) Number of patients with events and incidence

The order of description of risk names and risk names shall follow the e Sa sks, and in s definitions described in the Safety Specification (Important identified risks,

important potential risks, and important missing information).

# Case Summary for Post-marketing Surveillance, etc.

# Case summary in post-marketing surveillance, etc. (Attached Form 16)

Analysis Subjects evaluable for safety

population:

Analysis item: Case No.

Name of medical institution

Gender

Age

Reason for use (Disease code, disease name) Comorbidity (Disease code, disease name)

Route of administration

Maximum dose

Mean dose

Unit

Duration of use (duration of this drug treatment)

Concomitant medications (Drug code, drug name)

Degree of effect

Adverse reactions (Disease code, disease name, outcome)

CRF No.

Dropout

Reason for dropout

above analy.

"mination data entry
Notification No. 1119 (3) c
dated November 19, 2020. A list of the above analysis items will be prepared in accordance with the

reexamination data entry file preparation guideline specified in the

Notification No. 1119 (3) of the Pharmaceutical Evaluation Division, PSEHB

# **Preparation history (version control)**

| Version | Date | Author/Reporter | Comments |
|----------|-----------|-----------------|--------------------------------|
| Original | 2024 1 20 | | D C 1 |
| Version | 2024.1.30 | | Preparation of initial version |

Properly of Takeda, For non-commercial use only and subject to the applicable Temps of Use

# [Appendix 1] Comparison table of changes

| | | | After amendment Reason for change | |
|---|---|---|---|---|
| Page | Before amendment | After amendment | ~0°P1. | Reason for change |
| | | | 0,0, | |
| | | | HU | |
| | | | ) | |
| | | iec | | |
| | | enlo, | | |
| | | 29 | | |
| | | 31 | | |
| | | E.O. | | |
| | | Jus | | |
| | | , cilo | | |
| | ~ | 2 | | |
| | 201 | | | |
| | .000 | | | |
| | X 3/LC | | | |
| | Ex | 1 | | |
| | 6) | | | |
| 0,0 | Before amendment Before amendment Before amendment Before amendment | | | |
| X | | | | |